CLINICAL TRIAL: NCT01874678
Title: A Study of TS-1 Plus Cisplatin in Patients With Advanced Non-small-cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTYTG0904
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Non-small-cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TS-1/Cisplatin (Experimental): single arm
  Interventions: Drug: TS-1/Cisplatin

INTERVENTIONS:
Drug: TS-1/Cisplatin

SUMMARY:
Objectives:

1. Primary Objective:

   To bridge the data of efficacy in term of overall response rate of TS-1 plus cisplatin in Taiwanese advanced NSCLC patients from that gained from Japanese population
2. Secondary Objectives:

A. To assess progression free survival B. To assess overall survival C. To bridge the safety profile by assessing the toxicities and tolerability

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each subject must fulfill all of the following criteria:

1. histologically or cytologically confirmed non-small cell bronchogenic carcinoma
2. Stage IIIb or IV disease
3. presence of at least one measurable disease which is defined as lesion that can be measured in at least 1 dimension as ≥20 mm with conventional CT/MRI or ≥10 mm with spiral CT scan
4. performance status of ECOG 0, 1
5. age between 20 and 74 years at registration
6. life expectancy of at least 12 weeks
7. ability to take the oral study medication (TS-1)
8. voluntarily signed the written informed consent form.

Exclusion Criteria:

* other malignancy with the exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to the entry of study
* previously received chemotherapy or therapy with systemic anti-tumor effect
* significant co-morbid medical conditions, including, but not limited to , heart failure, renal failure, hepatic failure, hemorrhagic peptic ulcer, mechanical or paralytic ileus, or poorly controlled diabetes
* fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period and for three months following cessation of treatment
* Presence of mental disease or psychotic manifestation
* Participation in another clinical trial with any investigational drug within 30 days prior to entry
* judged ineligible by physicians for participation in the study due to safety concern.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
overall response rate | 2 year
  To assess overall response rate

SECONDARY OUTCOMES:
To assess progression free survival To assess overall survival To bridge the safety profile by assessing the toxicities and tolerability | 2 year
  To assess progression free survival To assess overall survival To bridge the safety profile by assessing the toxicities and tolerability

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Dalin Tzu Chi General Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Background] Okamoto I, Yoshioka H, Morita S, Ando M, Takeda K, Seto T, Yamamoto N, Saka H, Asami K, Hirashima T, Kudoh S, Satouchi M, Ikeda N, Iwamoto Y, Sawa T, Miyazaki M, Tamura K, Kurata T, Fukuoka M, Nakagawa K. Phase III trial comparing oral S-1 plus carboplatin with paclitaxel plus carboplatin in chemotherapy-naive patients with advanced non-small-cell lung cancer: results of a west Japan oncology group study. J Clin Oncol. 2010 Dec 20;28(36):5240-6. doi: 10.1200/JCO.2010.31.0326. Epub 2010 Nov 15. PMID 21079147
- [Background] Ichinose Y, Yoshimori K, Sakai H, Nakai Y, Sugiura T, Kawahara M, Niitani H. S-1 plus cisplatin combination chemotherapy in patients with advanced non-small cell lung cancer: a multi-institutional phase II trial. Clin Cancer Res. 2004 Dec 1;10(23):7860-4. doi: 10.1158/1078-0432.CCR-04-1200. PMID 15585618
- See also: TFDA — http://www.fda.gov.tw/TC/index.aspx